CLINICAL TRIAL: NCT03794999
Title: The Benralizumab Pregnancy Exposure Study: A VAMPSS Post Marketing Surveillance Study
Brief Title: Benralizumab Pregnancy Exposure Study
Status: Terminated | Type: Observational
Why Stopped: The decision to terminate the Fasenra pregnancy study and cancel the commitment to conduct additional pregnancy-related pharmacovigilance activities was made by the EMA following MAH's failed attempts to address patient recruitment challenges.
Sponsor: AstraZeneca (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: D3250R00026; EUPAS26461 (Registry Identifier: ENCePP)
Record Dates: First submitted 2018-12-04; First posted 2019-01-07 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Asthma
Keywords: asthma; pregnancy; benralizumab; infant; teratogenic
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Benralizumab-exposed group: Pregnant women with asthma exposed to benralizumab anytime during pregnancy or within 8 weeks prior to last menstrual period
  Interventions: Drug: Benralizumab-exposure
- Asthmatic comparison group: Pregnant women currently treated for asthma not exposed to benralizumab during pregnancy or within 8 weeks prior to last menstrual period
  Interventions: Drug: Exposure to other asthma medications
- Non-asthmatic comparison group: Pregnant women who are not diagnosed with asthma, have not had exposure to a known human teratogen, and have not taken benralizumab during pregnancy.

INTERVENTIONS:
Drug: Benralizumab-exposure — Exposure is defined as any dose of benralizumab for any length of time from 8 weeks prior to Last Mentrual Period (LMP) through the end of pregnancy, as reported by the mother and validated through medical record review. The 8-week cut-off prior to LMP is based upon the terminal half-life of benralizumab of approximately 15 days (clearance of benralizumab is based on five half-lives).
  Groups: Benralizumab-exposed group
Drug: Exposure to other asthma medications — Exposure to asthma medications for any number of days, at any dose, and at any time from LMP up to the date of enrollment, but no exposure to benralizumab during pregnancy or within 8 weeks prior to LMP.
  Groups: Asthmatic comparison group

SUMMARY:
This is a prospective, observational, exposure cohort study of pregnancy and infant outcomes in women with asthma exposed to benralizumab anytime during pregnancy, or within 8 weeks prior to the first day of the last menstrual period (LMP)

The objective of the study is to monitor planned or unplanned pregnancies to evaluate potential teratogenic effect (birth defect) when exposed to benralizumab compared to two unexposed comparator groups.

The primary outcome is major structural birth defects (abnormalities in development of structures of the body) and the secondary outcomes are preterm delivery (premature baby), small for gestational age infants (small for weight, length, and/or head circumference), spontaneous abortion (miscarriage), stillbirth (baby born without signs of life), elective termination (voluntary abortion) and small for age postnatal growth to one year of age (small for weight, length and/or head circumference). The birth prevalence or incidence of outcomes in women exposed to benralizumab, and their infants, will be compared to those observed in two unexposed comparator groups: a disease-matched comparison group of women who have not used benralizumab during pregnancy or within 8 weeks of their last menstrual period (LMP), but who have used other anti-asthmatic medications (treated disease comparison group), and a comparison group of healthy women who do not have a diagnosis of asthma, have not had exposure to a known human teratogen (substance that causes birth defect), and have not taken benralizumab in pregnancy (healthy comparison group).

ELIGIBILITY:
Participants will be recruited into the three cohorts concurrently, on the basis of the following inclusion/exclusion criteria:

Cohort 1: Benralizumab-Exposed

Inclusion Criteria:

* Currently pregnant women diagnosed with asthma who contact the OTIS Research Center and who have been exposed to benralizumab for any number of days, at any dose, and at any time from 8 weeks before the first day of LMP up to and including the end of pregnancy.
* Eligible participants will be currently pregnant women who agree to the conditions and requirements of the study including the interview schedule and release of medical records.

Exclusion Criteria:

* Women who have had exposure to another biologic, used for any indication, anytime during pregnancy or within 8 weeks of LMP.
* Women will not be eligible for Cohort 1 if they first contact the OTIS Research Center after prenatal diagnosis of a major structural birth defect.
* Restrospective cases (outcome of pregnancy known prior to enrollment).
* Women who have enrolled in the current study with a previous pregnancy.

Cohort 2: Treated Diseased Comparison

Inclusion Criteria:

* Currently pregnant women diagnosed with asthma and exposed to asthma medications for any number of days, at any dose, and at any time from LMP up to the date of enrollment, who contact the OTIS Research Center but who were not exposed to benralizumab during pregnancy or within 8 weeks prior to LMP.
* Eligible participants will be currently pregnant women who agree to the conditions and requirements of the study including the interview schedule and release of medical records.

Exclusion Criteria:

* Women with exposure to benralizumab any time during pregnancy or within 8 weeks prior to LMP.
* Women will not be eligible for Cohort 2 if they first come in contact with the OTIS Research Center after prenatal diagnosis of a major structural birth defect.
* Retrospective cases (outcome of pregnancy known prior to enrollment).
* Women who have enrolled in the current study with a previous pregnancy.

Cohort 3: Non-Asthmatic Comparison

Inclusion Criteria:

* Currently pregnant women who contact the OTIS Research Center.
* Eligible women may potentially have been exposed to non-teratogenic agents during this pregnancy.
* Women who agree to the conditions and requirements of the study including the interview schedule and release of medical records.

Exclusion Criteria:

* Women who have been exposed to any known teratogenic agents as determined by the OTIS Research Center (list in Annex 1) for any number of days, at any dose, from the first day of the last menstrual period up to and including the end of pregnancy.
* Women with a self-reported diagnosis of asthma, current or previous.
* Women will not be eligible for Cohort 3 if they come in contact with the OTIS Research Center after prenatal diagnosis of a major structural birth defect.
* Retrospective cases (outcome of pregnancy known prior to enrollment).
* Women who have enrolled in the current study with a previous pregnancy.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women who have or have not used benralizumab anytime in pregnancy for asthma.
Study Population: The study population includes pregnant women who reside in the US or Canada who have or have not used benralizumab anytime in pregnancy for asthma.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Major structural birth defects | Up to 1 year of age
  Pregnancies ending in live birth with exposure in the first trimester for benralizumab cohort, and other comparison groups at least one malformed infant in an individual pregnancy is considered one malformed outcome

SECONDARY OUTCOMES:
Spontaneous abortion/miscarriage | Prior to 20.0 weeks gestation
  Spontaneous pregnancy loss prior to 20.0 weeks gestation, since women only enrol after recognition of pregnancy, spontaneous abortions are only identified after enrolment in clinically recognised pregnancies.
Preterm delivery | Prior to 37 weeks of gestation
  Pregnancies enrolled prior to 37.0 weeks' gestation and ending in at least one live born infant. Excludes twins or higher order multiples due to inherent higher risk of preterm birth in multiples. Exposure can occur any time in pregnancy prior to the event.
Small for gestational age infants | At birth
  Pregnancies ending in at least one live born infant who are <10th centile on birth weight, length and/or head circumference for infant sex and gestational age; excluding twins or higher order multiples due to the inherent higher risk of reduced birth size in multiples. Exposure can occur any time in pregnancy prior to the event.
Stillbirth | At delivery
  Stillbirth is defined as a fetal death that occurs >20 weeks' gestation. All pregnancies, excluding lost-to-follow-up. Exposure can occur any time in pregnancy prior to the event.
Elective termination/abortion | At the end of pregnancy, or through 9 month pregnancy period
  Elective termination is defined as deliberate interruption of pregnancy by surgical or medical means. All pregnancies, excluding lost-to-follow-up. Exposure can occur anytime in pregnancy prior to the event.
Small for age postnatal growth of live born children to 1 year of age | Up to one year of age
  Postnatal growth is measured at approximately 1 year of age among live born infants and age and sex specific percentiles assigned using standard U.S. growth curves. Weight, length and/or head circumference <10th centile will be considered small for age. Multiples are excluded. Exposure can occur anytime in pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Chambers, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- Research Site, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00026&attachmentIdentifier=6ba559a5-7035-4629-90f4-a5ebcc42d2ed&fileName=OTIS_Benralizumab_Final_Analysis_Report_Synopsis_Redacted.pdf&versionIdentifier=